CLINICAL TRIAL: NCT01558921
Title: Randomized Multicentre Phase III Study of Short Course Radiation Therapy Followed by Prolonged Pre-operative Chemotherapy and Surgery in Primary High Risk Rectal Cancer Compared to Standard Chemoradiotherapy and Surgery and Optional Adjuvant Chemotherapy.
Brief Title: Rectal Cancer And Pre-operative Induction Therapy Followed by Dedicated Operation. The RAPIDO Trial
Acronym: RAPIDO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Karolinska University Hospital (Other); Leiden University Medical Center (Other); Uppsala University Hospital (Other); Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, B. van Etten, MD, PhD, Dr. B. van Etten, surgical oncologist, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL36315.042.11; 2010-023957-12 (EudraCT Number)
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; radiotherapy; chemotherapy; 5x5; capecitbine; oxaliplatin; CAPOX; FOLFOX; folinic acid; fluorouracil
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: standard arm: 5.5 weeks chemoradiation -> surgery -> optional chemotherapy experimental arm: 5x5Gy -> 12 wks chemotherapy -> surgery
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B: 5x5Gy -> CAPOX -> surgery (Experimental): experimental group (arm B) M1 scheme
  Interventions: Other: M1 scheme
- A: 5 weeks chemoradiation -> surgery (Active Comparator): control group (arm A) standard long course chemoradiotherapy
  Interventions: Other: standard long course chemoradiotherapy

INTERVENTIONS:
Other: M1 scheme — short course 5 x 5 Gy radiation scheme is followed by six cycles of combination chemotherapy (capecitabine and oxaliplatin (CAPOX)) and surgery. FOLFOX4 may be given as alternative for CAPOX
  Arms: B: 5x5Gy -> CAPOX -> surgery
Other: standard long course chemoradiotherapy — long course chemoradiotherapy followed by surgery. Optional adjuvant chemotherapy (CAPOX or FOLFOX) is allowed in the control group.
  Arms: A: 5 weeks chemoradiation -> surgery

SUMMARY:
Currently the 3-year disease free survival of patients with locally advanced rectal cancer is about 50%. Current standard treatment for patients at high risk of failing locally and/or systemically includes pre-operative long course radiotherapy (5 weeks) in combination with chemotherapy (so called neoadjuvant chemoradiotherapy). The neoadjuvant chemoradiotherapy has been demonstrated to improve local control, but had no effect on the overall survival. Different studies in patients with rectal cancer studying the effect of adjuvant post operative chemotherapy did not result in an improved survival. This may be due the fact that rectal cancer surgery (TME) is associated with a high complication rate so substantial proportion of patients cannot receive chemotherapy postoperatively. An alternative approach is to administer the systemic therapy preoperative. To guarantee control of the rectum tumor short-course radiotherapy (5 days) is given, as different studies showed local control of the tumor for a long time. During this waiting period the patient is in a good condition to receive an optimal dose of chemotherapy. The investigators hypothesize that with this proposed protocol both the local tumour and possible micrometastases are effectively treated and that this will result in an increased survival. The investigators will compare this with the standard treatment of neoadjuvant chemoradiation followed by TME surgery and optional adjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients will be randomized between an experimental group (arm B) in which short course 5 x 5 Gy radiation scheme is followed by six cycles of combination chemotherapy (capecitabine/5FU and oxaliplatin) and surgery and a control group (arm A) with long course chemoradiotherapy followed by surgery. In arm A adjuvant chemotherapy is allowed according to the local protocol of the institution. In both groups the rectal tumour will be removed by TME surgery or more extensive surgery if required because of tumour extent.

ELIGIBILITY:
Inclusion Criteria:

Primary tumour characteristics:

1. Histological proof of newly diagnosed primary adenocarcinoma of the rectum
2. Locally advanced tumour fulfilling at least one of the following criteria on pelvic MRI indicating high risk of failing locally and/or systemically (T4a, i.e. overgrowth to an adjacent organ or structure like the prostate, urinary bladder, uterus, sacrum, pelvic floor or side wall (according to TNM version 5), cT4b, i.e. peritoneal involvement, extramural vascular invasion (EMVI+). N2, i.e. four or more lymph nodes in the mesorectum showing morphological signs on MRI indicating metastatic disease. Positive MRF, i.e. tumor or lymph node < 1 mm from the mesorectal fascia. Enlarged lateral nodes, > 1 cm (lat LN+)

Exclusion Criteria:

1. Extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen
2. Presence of metastatic disease or recurrent rectal tumour
3. Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn¡¦s disease or active ulcerative Colitis
4. Concomitant malignancies, except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years
5. Known DPD deficiency
6. Any contraindications to MRI (e.g. patients with pacemakers)
7. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
8. Concurrent uncontrolled medical conditions
9. Any investigational treatment for rectal cancer within the past month
10. Pregnancy or breast feeding
11. Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract
12. Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia, e.g. atrial fibrillation, even if controlled with medication) or myocardial infarction within the past 12 months
13. Patients with symptoms or history of peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease related Treatment Failure (DrTF) | 3 year follow-up after surgery
  DrTF = Either local or distant relapse or death caused by the rectal carcinoma whichever comes first. In case of nonrectal cancer related death patients will be censored at date of death. In case of a second primary tumour patients will be censored at the date of diagnosis of the second primary tumour. In case of local regrowth after wait & watch strategy, followed by no resection or R2 resection, diagnosis local regrowth is taken. Patients lost to follow-up will be censored the last date of patient visit. Survival curves for Disease related Treatment Failure after 3 years of follow-up will be constructed using the method of Kaplan and Meier.

SECONDARY OUTCOMES:
Overall survival | 10 year
  Overall survival will be computed as the time between randomization and colorectal cancer or treatment related death. Patients lost to follow-up will be censored the last date of patient visit.
  In case of a second primary tumour patients will be censored at the date of diagnosis of the second primary tumour.
CRM negative rate | within 30 days
  Circumferential resection margin > 1 mm
pCR rate | within 30 days
  Pathological complete response after neo-adjuvant treatment
Short and long-term toxicity | 3 year follow-up
  Treatment associated toxicity
Surgical complications | 3 year follow-up
  Wound rupture, bleeding, infection, rectal anastomotic leak
Quality of life QLQ-C30 | 3 year after surgery
  Quality of life QLQ-C30
Quality of life QLQ-CR-29+ | 3 year after surgery
  Quality of life QLQ-CR-29+
Quality of life QLQ-CIPN20 | 3 year after surgery
  Quality of life QLQ-CIPN20
Quality of life LARS | 3 year after surgery
  LARS

CONTACTS AND LOCATIONS:
Overall Officials: B. van Etten, MD, PhD, Principal Investigator — University Medical Center Groningen, Department of Surgery, Groningen, The Netherlands; B. Glimelius, MD, PhD, Principal Investigator — Akademiska Sjukhuset, Department of Oncology, Uppsala, Sweden; G. A. Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen, Department of Medical Oncology, Groningen, The Netherlands; P. Nilsson, MD, PhD, Principal Investigator — Karolinska Universitetssjukhuset, Stockholm, Sweden; C. J. van de Velde, MD, PhD, Principal Investigator — Leiden University Medical Center, Department of Surgery, Leiden, The Netherlands; C.A.M. Marijnen, MD, PhD, Principal Investigator — Netherlands Cancer Institute, Amsterdam, the Netherlands
Locations (56):
- Siteman Cancer Center, Washington University Medical School, St Louis, Missouri, United States
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Odense Universitetshospital, Odense
- Netherlands (28):
  - University Medical Center Groningen, Groningen, PO BOX 30001
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, location VUMC, Amsterdam
  - Nki / Avl, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Deventer Hospital, Deventer
  - Catharina ZIekenhuis, Eindhoven
  - Het Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - de Tjongerschans, Heerenveen
  - Ziekenhuisgroep Twente, Hengelo
  - Spaarne Ziekenhuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Radiotherapeutisch Instituut Friesland, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - UMC Nijmegen St Radboud, Nijmegen
  - Antonius Ziekenhuis, Sneek
  - Bronovo Ziekenhuis, The Hague
  - HaGaZiekenhuis, The Hague
  - Medisch Centrum Haaglanden, The Hague
  - Diakonessenhuis, Utrecht
  - Isala Klinieken, Zwolle
- Norway (2):
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Oslo Universitetssykehus, Oslo
- Institute of Oncology, Ljubljana, Slovenia
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - ICO Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Consorcio Hospital General Universitario Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic la Fe, Valencia
- Sweden (17):
  - Södra Älvsborgs Sjukhus, Borås
  - Mälarsjukhuset, Eskilstuna
  - Falu Lasarett, Falun
  - Gävle sjukhus, Gävle
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Kalmar Hospital, Kalmar
  - Centralsjukhuset i Karlstad, Karlstad
  - Linköpings Universitet, Linköping
  - Universitetssjukhuset i Lund, Lund
  - Universitetssjukhuset ÖREBRO, Örebro
  - Skaraborgs Sjukhus, Skövde
  - Karolinska Universitetssjukhuset, Stockholm
  - Sundsvalls Sjukhus, Sundsvall
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
  - Centrallasarettet Växjö, Vaxjo
  - Centrallasarett, Västerås

REFERENCES:
- [Background] van der Valk MJM, Marijnen CAM, van Etten B, Dijkstra EA, Hilling DE, Kranenbarg EM, Putter H, Roodvoets AGH, Bahadoer RR, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes AMR, de Groot DJA, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; Collaborative investigators. Compliance and tolerability of short-course radiotherapy followed by preoperative chemotherapy and surgery for high-risk rectal cancer - Results of the international randomized RAPIDO-trial. Radiother Oncol. 2020 Jun;147:75-83. doi: 10.1016/j.radonc.2020.03.011. Epub 2020 Mar 30. PMID 32240909
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Background] Nilsson PJ, van Etten B, Hospers GA, Pahlman L, van de Velde CJ, Beets-Tan RG, Blomqvist L, Beukema JC, Kapiteijn E, Marijnen CA, Nagtegaal ID, Wiggers T, Glimelius B. Short-course radiotherapy followed by neo-adjuvant chemotherapy in locally advanced rectal cancer--the RAPIDO trial. BMC Cancer. 2013 Jun 7;13:279. doi: 10.1186/1471-2407-13-279. PMID 23742033
- [Background] Dijkstra EA, Hospers GAP, Kranenbarg EM, Fleer J, Roodvoets AGH, Bahadoer RR, Guren MG, Tjalma JJJ, Putter H, Crolla RMPH, Hendriks MP, Capdevila J, Radu C, van de Velde CJH, Nilsson PJ, Glimelius B, van Etten B, Marijnen CAM. Quality of life and late toxicity after short-course radiotherapy followed by chemotherapy or chemoradiotherapy for locally advanced rectal cancer - The RAPIDO trial. Radiother Oncol. 2022 Jun;171:69-76. doi: 10.1016/j.radonc.2022.04.013. Epub 2022 Apr 18. PMID 35447283
- [Background] Giunta EF, Bregni G, Pretta A, Deleporte A, Liberale G, Bali AM, Moretti L, Troiani T, Ciardiello F, Hendlisz A, Sclafani F. Total neoadjuvant therapy for rectal cancer: Making sense of the results from the RAPIDO and PRODIGE 23 trials. Cancer Treat Rev. 2021 May;96:102177. doi: 10.1016/j.ctrv.2021.102177. Epub 2021 Mar 16. PMID 33798955
- [Background] Jimenez-Fonseca P, Salazar R, Valenti V, Msaouel P, Carmona-Bayonas A. Is short-course radiotherapy and total neoadjuvant therapy the new standard of care in locally advanced rectal cancer? A sensitivity analysis of the RAPIDO clinical trial. Ann Oncol. 2022 Aug;33(8):786-793. doi: 10.1016/j.annonc.2022.04.010. Epub 2022 Apr 22. PMID 35462008
- [Background] Glynne-Jones R, Harrison M. Should the RAPIDO schedule represent standard of care in locally advanced rectal cancer? Ann Oncol. 2022 Aug;33(8):745-746. doi: 10.1016/j.annonc.2022.05.002. Epub 2022 May 12. No abstract available. PMID 35568280
- [Background] Patel A, Spychalski P, Corrao G, Jereczek-Fossa BA, Glynne-Jones R, Garcia-Aguilar J, Kobiela J. Neoadjuvant short-course radiotherapy with consolidation chemotherapy for locally advanced rectal cancer: a systematic review and meta-analysis. Acta Oncol. 2021 Oct;60(10):1308-1316. doi: 10.1080/0284186X.2021.1953137. Epub 2021 Jul 24. PMID 34308767
- [Background] Papaccio F, Rosello S, Huerta M, Gambardella V, Tarazona N, Fleitas T, Roda D, Cervantes A. Neoadjuvant Chemotherapy in Locally Advanced Rectal Cancer. Cancers (Basel). 2020 Dec 3;12(12):3611. doi: 10.3390/cancers12123611. PMID 33287114
- [Background] Dijkstra EA, Zwart WH, Putter H, Marijnen CAM, Nilsson PJ, van de Velde CJH, van Etten B, Hospers GAP, Glimelius B. Authors' reply-A sensitivity analysis of the RAPIDO clinical trial. Ann Oncol. 2023 Apr;34(4):446-447. doi: 10.1016/j.annonc.2022.12.012. Epub 2022 Dec 26. No abstract available. PMID 36581138
- See also: Dutch Colorectal CancerGroup — http://www.dccg.nl/trial/rapido

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT01558921/Prot_SAP_ICF_000.pdf